CLINICAL TRIAL: NCT05681234
Title: Clinical Application of 18F-labeled RD2 PET/CT Imaging in the Diagnosis and Treatment of Small Liver Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Principal Investigator, Chunjing Yu, Director, Affiliated Hospital of Jiangnan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LS2021058
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Liver Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-RD2 (Experimental)
  Interventions: Radiation: 18F-RD2

INTERVENTIONS:
Radiation: 18F-RD2 — Patients will receive 5-10 mCi 18F-RD2

SUMMARY:
This is a single arm study to evaluate the safety and biodistribution of 18F-labeled RD2 PET/CT Imaging in patients with small liver carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with highly suspected tumor；
2. Patients underwent PET/CT examination within 1 week;
3. Patients voluntarily signed informed consent;
4. Over 18 years old, male or female.

Exclusion Criteria:

1. Pregnant women;
2. Lactating women;
3. Patients with impaired renal function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of tissue distribution of 18F-RD2 | 2 hours
  Biodistribution of 18F-RD2 evaluated by radioactive uptake values (standardized uptake values, SUVs) in various organs during repeated 18F-RD2 scans will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China